CLINICAL TRIAL: NCT06320067
Title: Studying Treatments in Patients Receiving Androgen Deprivation Therapy (ADT) for Metastatic Prostate Cancer: Evaluation of Drug and Radiation Efficacy: A 2nd Multi-arm Multi-stage Randomised Controlled Trial (STAMPEDE2).
Brief Title: A Randomised Controlled Platform Trial Testing Treatments in Metastatic Hormone Sensitive Prostate Cancer
Acronym: STAMPEDE2
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University College, London (Other)
Collaborators: Cancer Research UK (Other); Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PR12; 1006437 (Other: IRAS)
Record Dates: First submitted 2024-01-10; First posted 2024-03-20 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Prostate Cancer Metastatic
Keywords: Hormone sensitive metastatic prostate cancer; Stereotactic ablative body radiotherapy (SABR); PSMA-Lutetium
MeSH Terms: interventions — Radiosurgery; Pluvicto; Lutetium; Lutetium-177; Androgen Antagonists; Docetaxel

STUDY DESIGN:
Intervention Model Description: Platform trial testing two research comparisons where patients are randomised either to experimental treatments in Arms S and P or their corresponding SoC control Arms A(S) and A(P).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Arm A of SABR Comparison (Active Comparator): SoC (ADT + ARPI ± docetaxel + local RT)
  Interventions: Drug: Androgen Deprivation Therapy (ADT); Drug: Androgen Receptor Signalling Inhibitor (ARPI); Radiation: Radiotherapy to Prostate ± Pelvic Nodes; Drug: Docetaxel
- Arm S of SABR Comparison (Experimental): SoC (ADT + ARPI ± docetaxel + local RT) + SABR
  Interventions: Radiation: Stereotactic Ablative Body Radiotherapy (SABR); Drug: Androgen Deprivation Therapy (ADT); Drug: Androgen Receptor Signalling Inhibitor (ARPI); Radiation: Radiotherapy to Prostate ± Pelvic Nodes; Drug: Docetaxel
- Arm A of 177Lu-PSMA-617 Comparison (Active Comparator): SoC (ADT + ARPI ± docetaxel ± local RT)
  Interventions: Drug: Androgen Deprivation Therapy (ADT); Drug: Androgen Receptor Signalling Inhibitor (ARPI); Radiation: Radiotherapy to Prostate ± Pelvic Nodes; Drug: Docetaxel
- Arm P of 177Lu-PSMA-617 Comparison (Experimental): SoC (ADT + ARPI ± docetaxel ± local RT) + 177Lu-PSMA-617
  Interventions: Other: 177Lu-PSMA-617; Drug: Androgen Deprivation Therapy (ADT); Drug: Androgen Receptor Signalling Inhibitor (ARPI); Radiation: Radiotherapy to Prostate ± Pelvic Nodes; Drug: Docetaxel

INTERVENTIONS:
Radiation: Stereotactic Ablative Body Radiotherapy (SABR) — SABR is a way of giving focused high-dose radiotherapy. SABR given with a dose fractionation schedule of 27-30Gy in 3-5 fractions over 1-2 weeks to up to 5 metastatic lesions in the bone and/or non-regional (extra-pelvic) lymph nodes.
  Other Names: Stereotactic body radiotherapy (SBRT)
  Arms: Arm S of SABR Comparison
Other: 177Lu-PSMA-617 — 177Lu-PSMA-617 is a nuclear medicine therapy. Patients will receive 177Lu-PSMA-617 to a dose of 7.4GBq. Each cycle will consist of 2 doses, 1 week apart (on day 1 and day 8) and will last 6 weeks. Treatment will be given for up to 3 cycles (6 doses).
  Other Names: Lutetium (177Lu) Vipivotide Tetraxetan; AAA617; Pluvicto
  Arms: Arm P of 177Lu-PSMA-617 Comparison
Drug: Androgen Deprivation Therapy (ADT) — Long-term, continuous treatment with ADT (bilateral orchidectomy, LHRH agonists or LHRH antagonists) if not previously surgically castrated. The choice of ADT is at the discretion of the investigator. This will be given as standard of care as per local guidelines.
Drug: Androgen Receptor Signalling Inhibitor (ARPI) — Second generation ARPI (Abiraterone Acetate and Prednisolone, Enzalutamide, Apalutamide or Darolutamide). This will be given as standard of care as per local guidelines.
  Abiraterone acetate will be administered as a single 1000mg once daily dose (4 tablets to be taken together once a day) with prednisolone 5mg once daily to prevent secondary mineralocorticoid excess.
  Enzalutamide will be administered as a 160mg oral dose (four capsules taken together at the same time every day) with or without food. Enzalutamide is administered daily in 28-day cycles.
  Apalutamide will be administered as 240mg oral dose (four tablets taken together at the same time every day) with or without food. Apalutamide is administered daily in 28-day cycles. Patients require thyroid function monitoring.
  Darolutamide will be administered as 600mg oral dose (two 300mg tablets taken together) with or without food. Darolutamide is administered twice daily in 28-day cycles.
Radiation: Radiotherapy to Prostate ± Pelvic Nodes — Either 36.25Gy given in 5 fractions over 1-2 weeks to prostate or 60Gy in 20 fractions over 4 weeks to prostate (± 44-47Gy in 20 fractions to pelvic lymph nodes ± 51Gy in 20 fractions boost to involved nodes).
Drug: Docetaxel — Maximum of 6 cycles every 3 weeks may be given at a dose of 75mg/m2 by IV infusion.

SUMMARY:
STAMPEDE2 is a clinical trial comparing two new treatments with standard of care in people with prostate cancer that has spread to other parts of the body and is responsive to hormone therapy. People from all backgrounds and ethnicities are encouraged to take part and multiple hospitals across the UK are involved. University College London is running the trial.

Each comparison within the trial has its own control arm where people get the best standard of care (Arm A) versus a research arm where a new treatment is added to standard of care.

Participants are allocated to an arm by a computerised system with a 50% chance of getting the research treatment.

Comparison S: Arm A versus Arm S (Stereotactic Ablative Body Radiotherapy (SABR)) - Tests whether giving targeted doses of radiotherapy (SABR) to parts of the body where the cancer has spread slows the spread of the cancer and improves survival. 2476 people will be in this comparison.

Comparison P: Arm A versus Arm P (PSMA-Lutetium (177Lu-PSMA-617)) - Tests whether giving a radioactive material (177Lu-PSMA-617) that targets prostate cancer cells slows the spread of the cancer and improves survival. 1756 people will be in this comparison.

All participants will be followed up with scans and tests to monitor their cancer. Doctors will check for any side effects from the treatments. Treatments will be stopped if side effects are serious, or people no longer wish to take the treatments.

ELIGIBILITY:
Registration Inclusion Criteria:

1. At least 18 years old.
2. Histological confirmation of prostate adenocarcinoma or a strong clinical suspicion of prostate cancer with a plan to confirm the diagnosis formally before any future randomisation.
3. Confirmation of metastatic site(s) on CT/MRI and either bone or PET scan. Patients with metastatic disease meeting any of the following criteria are eligible:

   * Metastatic disease to the bone (in any distribution).
   * Non-regional lymph node metastases of any size or distribution. Lymph nodes that are only visible on PET will not be eligible as sites of metastasis. Note: If lymph nodes are the only site of metastases, then at least one must be at least 1.5cm in short axis AND outside of the pelvis.
   * Visceral metastases of any size or distribution.
4. Clinical presentation is:

   A. de novo. OR B. relapsed with; (1) continuing hormone sensitivity in the opinion of the investigator, and; (2) all hormone treatments (e.g., ADT and ARPI) will have been completed ≥2 years prior to any future randomisation into any of the comparisons, and; (3) will have received ≤3 years total of ADT at the point of randomisation into any comparison.

   Note: the dates will be checked again at randomisation. It is the responsibility of the investigator to account for the time between registration and randomisation into any comparison.
5. Long-term androgen deprivation therapy (ADT) has started or there is an intention to start for a minimum of 2 years.
6. WHO Performance Status 0-2 or, if WHO Performance Status 3, deemed to be due to metastatic burden and expected to improve with ADT. Note: Improvement to WHO status 0-2 will be checked again at randomisation into any subsequent comparison.

   Note: For WHO performance status definitions see Appendix 1.
7. Willing and able to comply with trial treatments.
8. Patient has signed informed consent form for registration into the STAMPEDE2 Trial platform.

Registration Exclusion Criteria:

1. Clinically and pathologically overt small cell carcinoma.
2. Metastatic brain disease or leptomeningeal disease.
3. Any active malignancies (i.e., progressing or requiring any treatment in the previous 36 months) other than prostate cancer (except non-muscle invasive bladder cancer; nonmelanomatous skin cancer or a malignancy that is considered cured with minimal risk of recurrence).
4. Any other medical condition that in the investigator's opinion means the participant is unfit or unsuitable for long-term ADT or the trial treatments in the comparison for which they are being considered.

Eligibility Criteria For Comparison S Testing SABR:

Patients who meet the general eligibility criteria can be considered for the SABR comparison. Recruiting sites will assess metastatic disease burden using CT/MRI scans and baseline Tc-99m bone scan or PET scan to assess number of metastatic bone and non-regional lymph node foci, and presence of visceral metastases. Patients will be classified as either 'SABR-eligible' or 'SABR-ineligible' using the following definition.

Definition of SABR-eligible disease:

Patients will be classified as SABR-eligible if they meet all the following criteria:

* 1-5 metastatic lesions (including either bone and/or non-regional lymph node sites).
* Clinician determination that metastatic lesions are considered suitable for SABR on technical grounds (such as proximity of dose limiting normal tissue or tumour volume). Note: Clinical determination can consider next-generation imaging (e.g., PSMA PET-CT or WBMRI) where available. It is the investigator's responsibility to consider the impact of any findings on the suitability of SABR for the patient. Any next-generation imaging used prior to randomisation should be declared at randomisation so that it can be used as a stratification factor.
* Absence of visceral metastases.

Otherwise, patients will be classified as SABR-ineligible.

In addition to the general registration eligibility criteria, they need to meet all the following criteria for entry into Comparison S:

1. Patient still meets all eligibility criteria for registration in Section 4.4.
2. Histological confirmation of prostate adenocarcinoma.
3. Newly diagnosed (de novo) metastatic disease that is considered eligible for SABR according to the above definition.
4. Patient has started ADT and randomisation is ≤12 weeks since the start of ADT.
5. WHO performance status 0-2 (see Appendix 1).
6. Patient has provided signed informed consent for participation in Comparison S.

Exclusion Criteria For Comparison S Testing SABR:

1. Patient has relapsed prostate cancer.
2. Prior radical treatment to the prostate (e.g., radical surgery and/or radiotherapy).
3. Intracranial metastatic disease.
4. Prior treatment to a metastatic site (e.g., radiotherapy, surgery or RFA).
5. Significant or progressive neurological deficit such that emergency (within 24 hours) surgery or radiation required (e.g., metastatic spinal cord compression, or impingement of the cord or any other clinical scenario whereby urgent radiotherapy to the spine is required).
6. Any condition or co-morbidities that, in the judgement of the clinician, preclude procedures required to facilitate radiotherapy delivery e.g.:

   1. Disease staging and follow-up.
   2. Radiotherapy planning procedures.
7. Any condition or co-morbidities that, in the judgement of the clinician, preclude the safe delivery of radiotherapy to the prostate (± pelvic lymph nodes) and/or metastases e.g., inflammatory bowel disease, significant systemic connective tissue disorder, radiological evidence of idiopathic pulmonary fibrosis).
8. Active malignancy other than prostate cancer within the last 36 months.

Eligibility Criteria For Comparison P Testing 177LU-PSMA-617:

In addition to the general eligibility criteria, patients need to meet the following criteria for entry into Comparison P:

1. Patient still meets all eligibility criteria for registration.
2. Histological confirmation of prostate adenocarcinoma.
3. Patient meets the definition of SABR ineligible disease.
4. Patients must have adequate organ function as indicated by blood tests within 4 weeks prior to randomisation:

   Bone marrow function
   1. ANC ≥1.5 x 109/L
   2. Platelets ≥100 x 109/L
   3. Haemoglobin ≥9g/dL, independent of transfusions for at least 28 days Hepatic function

   <!-- -->

   1. Total bilirubin ≤2 x ULN. For patients with Gilbert's Syndrome ≤3 x ULN is permitted.
   2. AST and/or ALT performed with all results ≤3 × ULN or ≤5 x ULN for patients with liver metastasis Renal Function

   <!-- -->

   1. EGFR ≥50 mL/min/1.73m2 calculated using the MDRD formula
   2. Albumin ≥25g/L
5. Patient has started ADT and randomisation is ≤12 weeks since start of current ADT.
6. If relapsed disease, prior LHRH agonist/antagonist with or without first generation antiandrogen use in the adjuvant/neo-adjuvant setting, hormone treatment must have been discontinued ≥2 years prior to randomisation AND must not have exceeded a total of >3 years of therapy AND must not have shown disease progression within 12 months of completing adjuvant/neo-adjuvant therapy.
7. WHO performance status 0-2 (see Appendix 1).
8. Patient has provided signed informed consent for participation in Comparison P.

Exclusion Criteria For Comparison P Testing 177Lu-PSMA-617:

1. Prior treatment with any of the following:

   1. Strontium-89, Samarium-153, Rhenium-186, Rhenium-188, Radium-223
   2. PSMA-targeted radioligand therapy
2. Symptomatic cord compression, or clinical/radiological findings indicative of impending cord compression.
3. Any condition that precludes raised arms position.
4. Unmanageable bladder outflow obstruction or urinary incontinence. Note: bladder outflow obstruction or urinary incontinence which is manageable and controlled with best available standard of care (incl. drainage, pads) is permitted.
5. Imaging Sub-study only: Contraindication to MRI (e.g., pacemakers, except MRI compatible pacemakers).

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3360 (Estimated)
Dates: Start 2024-06-11 (Actual); Primary Completion 2031-04 (Estimated); Study Completion 2032-03 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS) | Final analysis for each comparison triggered when adequate number of death events have occurred in control arm of each comparison. Anticipate final reporting for OS in Comparison S: ~84 months (7 years) from FPFV, P: ~64 months (5.3 years) from FPFV.
  OS is defined as time from randomisation to death from any cause.
  The final reporting times of OS for each comparison below will depend on the recruitment rates and the accuracy of assumed median survival times in the sample size calculations.

SECONDARY OUTCOMES:
Failure-Free Survival (FFS) | Up to 10 years from randomisation. FFS is declared as a secondary outcome and is not part of sample size calculations, nor timelines for the study.
  Time from randomisation until the first of:
  * Biochemical progression
  * Clinical progression such as symptomatic local progression leading to intervention
  * Radiographic confirmed progression including local progression, pelvic lymph node progression, progression of an existing metastatic site or development of new metastatic site defined as lymph nodes outside the pelvis, bone or organ involvement
  * Symptomatic skeletal-related events secondary to cancer progression
  * Death from any cause
Radiographic Progression-Free-Survival (rPFS) | Up to 10 years from randomisation. rPFS is declared as a secondary outcome and is not part of sample size calculations, nor timelines for the study.
  Time from randomisation until the first of:
  * Radiographic confirmed progression of an existing metastatic site or development of a new metastatic site defined as lymph nodes outside the pelvis, bone or organ involvement
  * Symptomatic skeletal-related events secondary to cancer progression
  * Death from any cause
Prostate cancer specific survival (PCSS) | Up to 10 years from randomisation. PCSS is declared as a secondary outcome and is not part of the sample size calculations, nor timelines for the study.
  Time from randomisation to death from prostate cancer.
Safety through reporting of SAEs | S: until 6 months after randomisation; P: until 6 months after randomisation or 40 days after completion or permanent discontinuation of an IMP 177Lu-PSMA-617 (whichever is furthest); N: until 30 days after permanent discontinuation of an IMP
Toxicity using CTCAE classification and reporting of all Adverse Events that are ≥ grade 3 or grade 1 and 2 leading to a change in trial treatment | All safety and toxicity data will be presented by randomised group. The exact nature of this will be pre-specified in the statistical analysis plan that is still in development.
Compliance with randomised allocation. Formal definitions for compliance with treatment will be pre-specified in the statistical analysis plan. This is still in development. | Randomisation until death or end of trial treatment (up to 10 years from randomisation).
Resource use for cost-effectiveness assessment | Randomisation until death or end of trial treatment (up to 10 years from randomisation).
EQ-5D-5L questionnaire for QoL and cost effectiveness assessment | From date of randomisation until death or end of trial, whichever came first (up to 10 years from randomisation). The end of the trial will be determined by the timelines described in the primary outcomes section.

CONTACTS AND LOCATIONS:
Overall Officials: Louise Brown, Study Director — MRC CTU at UCL; Nick James, Principal Investigator — Institute of Cancer Research, United Kingdom
Locations (18):
- United Kingdom (18):
  - Mount Vernon Hospital, Barnsley
  - Addenbrookes, Cambridge
  - Royal Devon University Hospital Trust, Exeter
  - Royal Devon & Exeter Hospital, Exeter
  - The Princess Alexandra Hospital, Harlow
  - University College London Hospitals NHS Foundation Trust, London
  - The Royal Marsden Hospital, London
  - Barts Health NHS Trust, London
  - North Middlesex Hospital, London
  - Royal Free Hospital, London
  - The James Cook University Hospital, Middlesbrough
  - Churchill Hospital, Oxford
  - Derriford Hospital, Plymouth
  - Queen Alexandra Hospital, Portsmouth
  - Barking, Havering and Redbridge University Hospitals NHS Trust, Romford
  - North Tees Health NHS Trust, Stockton-on-Tees
  - The Royal Marsden Hospital, Sutton
  - Kings Mill Hospital, Sutton in Ashfield

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared according to the CTU's controlled access approach based on principles outlined in the trial protocol.
  Requests for sharing data will need to provide detail on the specific requirements, proposed research, qualifications of researchers and publication plan. All non-identifiable data will be available for sharing if approved following the CTU review process. Access to the digital image repository and the stored pathological tissue from researchers outside of the MRC CTU will be obtained through a formal data sharing application detailing the specific requirements, proposed research, investigator qualifications and publication plan. Applications for access to tissue are required separately from access to the shared clinical data.
Supporting Information: Study Protocol
Time Frame: It will become available for data sharing requests through the MRC CTU process following the primary analysis publication. Research data will be stored a minimum of 25 years.
Access Criteria: Data will be available for sharing and researchers wishing to access STAMPEDE2 data should contact the Trial Management Group via the CTU Trial team using the study mailbox in the first instance.
  A formal data sharing process has been developed at the MRC CTU. Requests for sharing data will need to provide detail on the specific requirements, proposed research, qualifications of researchers and publication plan. The requests will be reviewed by the appropriate STAMPEDE2 committees. A data transfer agreement will be signed prior to the transfer of any information. All patients will be consented for future data sharing and if data requests are approved, only anonymised data will be sent using appropriately encrypted methods for data transfer.

REFERENCES:
- See also: Related Info — http://www.stampede2trial.org